CLINICAL TRIAL: NCT02816073
Title: Single-session Pattern Scanning Laser Pan-retinal Photocoagulation in Proliferative Diabetic Retinopathy - a Randomized Study
Brief Title: Pattern Scanning Laser Pan-retinal Photocoagulation in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Christian Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung-yee Chung, Associate Consultant, United Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0079
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Retinopathy; Lasers; Treatment Outcome
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1,700 (Active Comparator): Patients receive 1,700 (+/- 5%) laser shots in a single session of pan-retinal photocoagulation using pattern scanning laser
  Interventions: Device: Pan-retinal photocoagulation using pattern scanning laser
- 2,500 (Active Comparator): Patients receive 2,500 (+/- 5%) laser shots in a single session of pan-retinal photocoagulation using pattern scanning laser
  Interventions: Device: Pan-retinal photocoagulation using pattern scanning laser

INTERVENTIONS:
Device: Pan-retinal photocoagulation using pattern scanning laser — Patients receive the designated number of laser shots of pan-retinal photocoagulation with pattern scanning laser in a single session

SUMMARY:
A randomized study to assess the safety and efficacy of single-session pan-retinal photocoagulation (PRP) using Pattern Scan Laser (PASCAL) in proliferative diabetic retinopathy (PDR) - 1,700 shots vs 2,500 shots

ELIGIBILITY:
Inclusion Criteria:

* All treatment-naïve patients with proliferative diabetic retinopathy (PDR) who attended our ophthalmic clinic from 1st December 2012 to 30th November

Exclusion Criteria:

* significant media opacity affecting laser uptake (e.g. corneal opacity, mature cataract, dense vitreous haemorrhage)
* any pre-existing ocular disorders resulting in visual impairment (e.g. retinal degenerations, maculopathies, primary glaucoma and other optic neuropathies)
* those who received previous retinal laser treatment, intravitreal injections or intraocular surgeries
* clinically significant macular oedema on clinical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Regression of neovascularization | 3 months
  Fluorescein angiogram assessment by independent observer

SECONDARY OUTCOMES:
Activity of neovascularization | 3 months
  Descriptive analysis of fundus fluorescein angiogram by independent observer into 4 categories: no leakage, reduced leakage, same leakage, increased leakage
Best corrected visual acuity | 1 week, 1 month, 3 months, 6 months
Complications | 1 week, 1 month, 3 months, 6 months
  choroidal detachment, exudative retinal detachment, retinal breaks
Central foveal thickness | 1 week
  Measured by spectral domain optical coherence tomography (Heidelberg Spectralis)
Retreatment rate | 6 months
  Patients requiring retreatment with pan-retinal photocoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth KW Li, MBChB, Principal Investigator — United Christian Hospital; The University of Hong Kong